CLINICAL TRIAL: NCT03156361
Title: A Randomized Controlled Trial Comparing 21 Days of Continuous Subcutaneous Insulin Infusion (CSII) Using Hepatic Directed Vesicle (HDV) Insulin to Standard CSII in Type 1 Diabetes Mellitus
Brief Title: 21 Day Comparison of Continuous Insulin Infusion Using HDV Insulin to Standard Insulin in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diasome Pharmaceuticals (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP 01-2017-02
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2017-04

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Intervention Model Description: This is a single center, double blind, active comparator controlled 2-Way crossover multiple dose safety, tolerability and efficacy study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HDV insulin lispro 100 UNIT/mL (Experimental): Hepatic Directed Vesicle (HDV) is the active excipient, added to insulin lispro. HDV binds to a portion of the insulin lispro.
  Interventions: Drug: HDV insulin lispro 100 UNIT/mL
- Insulin Lispro 100 UNIT/mL (Active Comparator): Sterile Water for Injection (SWFI) is added to the insulin lispro, to dilute the insulin lispro equal to the HDV insulin lispro
  Interventions: Drug: Insulin Lispro 100 Units/mL

INTERVENTIONS:
Drug: HDV insulin lispro 100 UNIT/mL — Hepatic Directed Vesicle (HDV) added to commercial insulin lispro
  Other Names: HDV Humalog
  Arms: HDV insulin lispro 100 UNIT/mL
Drug: Insulin Lispro 100 Units/mL — Sterile Water for Injection added to commercial insulin lispro
  Other Names: Humalog
  Arms: Insulin Lispro 100 UNIT/mL

SUMMARY:
Single Center, Double Blind, Active Comparator Controlled 2-Way Crossover Multiple Dose Safety, Tolerability and Efficacy Study

DETAILED DESCRIPTION:
This is a single center, double blind, active comparator controlled 2-Way crossover multiple dose safety, tolerability and efficacy study.

The study will consist of three periods. Total duration will be approximately nine weeks, including a screening period of up to 14 days, a 7-day run-in period and two 21-day treatment periods.

Subjects will be screened and then they will undergo a week of baseline CGM. They will then be randomized to one of two treatment sequences: three weeks of treatment with HDV-lispro followed by three weeks of treatment with insulin lispro diluted with sterile water to match the insulin concentration in HDV-lispro, or the same treatments in the reverse order.

A test meal study (standardized liquid test meal) is to be conducted at the beginning of treatment (baseline study) and at the end of each three week treatment period. As noted above, frequent blood samples will be collected for glucose and insulin levels during the first (baseline study) test meal; during the two test meals performed after the two treatment periods the same sampling for glucose and insulin will be performed, with the addition of collecting samples for glucagon levels.

Subjects will also perform blinded continuous glucose monitoring throughout the entirety of the study (7 weeks).

Throughout study, subjects will be asked to perform frequent self-monitoring of blood glucose (SMBG), at least 6 times per day (before and 60-90 minutes after each meal) during 3 or more days of each week. This will serve as data for therapeutic decision-making as well as for data collection.

ELIGIBILITY:
Inclusion Criteria:

1. T1DM ≥12 months
2. C-peptide <0.6 ng/mL (a single re-test is allowable)
3. Treatment with rapid analog insulin by CSII for the previous 6 months
4. Familiarity with continuous glucose monitoring (CGM) technology; subjects nee d not be currently using CGM but should have used it in the past. Personal (unblinded) CGM will NOT be allowed during the study
5. Willingness to use insulin lispro as the analog insulin during the study period
6. Use of MiniMed Paradigm® pump for the previous 6 months. Pumps that employ low glucose suspend technology will NOT be allowed during the study
7. BMI ≥18.0 kg/m2 and ≤35.0 kg/m2
8. A1C≤9.0% (a single re-test is allowable)

Exclusion Criteria:

1. Known or suspected allergy to any component of any of the study drugs in this trial.
2. A patient who has unstable proliferative retinopathy or maculopathy, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
3. Use of oral anti-diabetic or non-insulin anti-diabetic injection therapies (e.g. SGLT-2 inhibitors, pramlintide, GLP-1 agonists, etc.)
4. Current smokers; if a former smoker, no tobacco products (inhaled, oral or buccal) for the previous 3 months
5. As judged by the investigator, clinically significant active disease of the gastrointestinal, cardiovascular (including a history of arrhythmia or conduction delays on ECG), hepatic, neurological, renal, genitourinary, or hematological systems, or uncontrolled hypertension (diastolic blood pressure ≥ 100 mmHg and/or systolic blood pressure ≥ 160 mmHg after 5 minutes in the supine position).
6. History of any illness or disease that in the opinion of the Investigator might confound the results of the trial or pose additional risk in administering the study drugs to the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Glucose area under the curve | 21 days
  To evaluate glucose response (incremental AUC) to standardized test meal challenge following 21 days of CSII treatment with HDV insulin lispro versus insulin lispro diluted with sterile water

SECONDARY OUTCOMES:
total units Insulin | 21 days
  To compare insulin doses (basal, bolus and total) during HDV insulin lispro treatment

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Muchmore, MD, Study Director — Diasome Pharmaceuticals
Locations (1):
- Atlanta Diabetes Association, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No